CLINICAL TRIAL: NCT06032871
Title: Comparison of Two Airway Clearance Techniques by Electrical Impedance Tomography- a Parallel Study
Brief Title: Comparisons of Two Airway Clearance Techniques
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hui-Ling Lin (Other)
Responsible Party: Sponsor-Investigator, Hui-Ling Lin, Professor, Chang Gung University
Organization: Chang Gung University (Other)
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Supportive Care
Other Study IDs: IRB2212210081
Record Dates: First submitted 2023-09-05; First posted 2023-09-13 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: Airway Clearance Impairment
Keywords: Airway clearance technique; Ventilator associated pneumonia; Electrical impedance tomography; High frequency chest wall oscillation; Chest physiotherapy
MeSH Terms: conditions — Pneumonia, Ventilator-Associated | interventions — Chest Wall Oscillation

STUDY DESIGN:
Masking Description: The group will be coded and masked to the investigator and the outcome accessor.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Chest physiotherapy (Experimental): Patients receive airway clearance by chest physiotherapy for 30 minutes twice a day.
  Interventions: Procedure: Chest physiotherapy
- High frequency chest wall oscillation (Experimental): Participants received high frequency chest wall oscillation therapy twice a dy
  Interventions: Procedure: high frequency chest wall oscillation

INTERVENTIONS:
Procedure: high frequency chest wall oscillation — Patients receive airway clearance by high frequency chest wall oscillation for 30 minutes twice a day.
  Arms: High frequency chest wall oscillation
Procedure: Chest physiotherapy — Participants received chest physiotherapy twice a day
  Arms: Chest physiotherapy

SUMMARY:
The goal of this clinical trial is to compare the effectiveness of two airway clearance techniques for patients with ventilator associated pneumonia. The main questions it aim to answer are:

* effect of the therapies on volume changes
* outcome on sputum clearance Participants will receive airway clearance techniques of
* chest physiotherapy
* high frequency chest wall oscillation.

DETAILED DESCRIPTION:
Sputum can be accumulated in the airways of intubated patients, resulting in recurrent pneumonia. The airway clearance therapy is often utilized with chest physiotherapy or high frequency chest wall oscillation which has become popular for its easy of use and less time consuming to the healthcare workers. The main questions it aim to answer are on effectiveness of the therapies on lung volume changes and sputum clearance by two airway clearance techniques. With the oscillation of entire chest wall, the investigators hypothesize that the high frequency chest wall oscillation is more effectively clear sputum in the distal airways.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with chronic pulmonary disease
* Diagnosed with ventilator associated pneumonia
* Receive airway clearance therapy

Exclusion Criteria:

* Head injury, spinal injury
* Instable hemodynamics
* Intercranial pressure > 20 cmH2O
* Active hemoptysis
* Empyema
* Eye surgery
* Abdominal distension
* Chest tube insertion
* Active tuberculosis

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2023-03-16 (Actual); Primary Completion 2023-12-12 (Actual); Study Completion 2023-12-30 (Actual)

PRIMARY OUTCOMES:
end-expiratory lung impedance | Measurement before intervention, 30 after, 1 hour and 2 hours after intervention
  Changes of global of impedance of lungs measure by the electrical impedance tomography

SECONDARY OUTCOMES:
Weight of secretions | Sputum is collected before intervention, 30 after, 1 hour and 2 hours after intervention
  Sputum amount is weighted.

CONTACTS AND LOCATIONS:
Overall Officials: Hui-Ling Lin, PhD, Principal Investigator — Chang Gung University
Locations (2):
- Taiwan (2):
  - Linkou Chang Gung Memorial Hospital, Taoyuan District
  - Chang Gung Memorial Hospital, Taoyuan District

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Rowley DD, Malinowski TP, Di Peppe JL, Sharkey RM, Gochenour DU, Enfield KB. A Randomized Controlled Trial Comparing Two Lung Expansion Therapies After Upper Abdominal Surgery. Respir Care. 2019 Oct;64(10):1181-1192. doi: 10.4187/respcare.06812. Epub 2019 May 21. PMID 31113857